CLINICAL TRIAL: NCT03141645
Title: Comparison of Preoperative Intravenous Fluid Loading and Ondansetron in Reduction of Incidence Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy: A Prospective Randomized Controlled Study
Brief Title: Comparison of IV Fluid Loading and Ondansetron in Reduction of PONV After LC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Collaborators: Buddhachinaraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Assistant Professor, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SIRB007
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Nausea; Postoperative Vomiting; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fluid loading group (Experimental): Patients will receive ringer lactate solution 10ml/kg in 15 minutes before starting operation
  Interventions: Other: Fluid loading
- Ondansetron group (Active Comparator): Patients will receive an 8 mg of intravenous ondansetron in 15 minutes before finishing operation.
  Interventions: Drug: Ondansetron
- Control group (No Intervention): Patients will receive neither preoperative intravenous fluid loading nor intravenous ondansetron.

INTERVENTIONS:
Other: Fluid loading — Patients in the preoperative intravenous fluid loading group (group F) will receive ringer lactate solution 10ml/kg in 15 minutes before starting operation.
  Other Names: Preoperative IV loading
  Arms: Fluid loading group
Drug: Ondansetron — Patients in the ondansetron group (group O) will receive an 8 mg of intravenous ondansetron in 15 minutes before finishing operation
  Other Names: Zetron
  Arms: Ondansetron group

SUMMARY:
This study is designed to examine the incidence of postoperative nausea and vomiting during 24 hours after elective laparoscopic cholecystectomy in patients receiving preoperative intravenous fluid loading (group F), ondansetron (group O) and receiving neither fluid nor ondansetron or control group (group C).

DETAILED DESCRIPTION:
This study is a prospective randomized control trial. It is designed to examine the incidence of postoperative nausea and vomiting during 24 hours after elective laparoscopic cholecystectomy in patients receiving preoperative intravenous fluid loading (group F), ondansetron (group O) and receiving neither fluid nor ondansetron or control group (group C). This study is hypothesized that the incidence of PONV in patients receiving preoperative intravenous fluid loading (group F) and patients receiving ondansetron (group O) will be similarly reduced from the control group (receiving neither fluid nor ondansetron).

ELIGIBILITY:
Inclusion Criteria:

* patients with aged 18 to 70 years with an ASA physical status 1-3

Exclusion Criteria including patients

* with pregnant or breast-feeding patients
* having history of taking antiemetic drugs within 24 hours before surgery
* with hypersensitivity or allergy to ondansetron
* with CKD stage 4, 5
* with congestive heart failure, LVEF <40
* with cirrhosis child c
* refusal or cannot communicate or understand the purpose of this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative nausea and vomiting | 24 hours
  The incidence of postoperative nausea and vomiting within postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, MD, MSc, Principal Investigator — Faculty of Medicine Siririaj Hospital
Locations (1):
- Mingkwan Wongyingsinn, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wongyingsinn M, Peanpanich P, Charoensawan S. A randomized controlled trial comparing incidences of postoperative nausea and vomiting after laparoscopic cholecystectomy for preoperative intravenous fluid loading, ondansetron, and control groups in a regional hospital setting in a developing country. Medicine (Baltimore). 2022 Oct 21;101(42):e31155. doi: 10.1097/MD.0000000000031155. PMID 36281094